CLINICAL TRIAL: NCT05171088
Title: Colorectal Resection in Emergency General Surgery - To Anastomose, or Not to Anastomose
Brief Title: Colorectal Resection in Emergency General Surgery
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 100.GME.2018.D
Record Dates: First submitted 2020-11-18; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Resection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary anastomosis is associated with higher rates of perioperative morbidity/mortality and that fecal diversion improves overall mortality, decreases length of stay, and lowers rates of surgical complications requiring unplanned operative intervention.

DETAILED DESCRIPTION:
This is a prospective observational study. All patients undergoing colon resection in the urgent/emergent setting meeting our inclusion/exclusion criteria will be enrolled in the study. Data will be collected prospectively and the decision to perform proximal diversion or anastomosis is solely the responsibility of the managing acute care surgeon. No guidelines or protocols will be suggested so as to avoid any influence on practitioner decision-making. The plan is to complete the data collection and analysis by 03/01/2020

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing urgent/emergent colon resection (less than 24 hours after decision to operate) by an acute care surgeon

Exclusion Criteria:

* Elective operations performed by acute care surgeons within 24-hours of the decision to operate (e.g., scheduled resection of non-obstructed, non-perforated malignancy)
* Prisoners
* Pregnancy
* Wards of the state
* Patients less than 18-years of age
* Traumatic mechanisms of injury
* Death within 24-hours of index operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing colon resection at Methodist Dallas Medical Center in the urgent/emergent setting meeting our inclusion/exclusion criteria will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Perioperative mortality and need for unplanned procedural intervention | 1 days to 12 months
  Perioperative mortality and need for unplanned procedural intervention (intervention by a surgeon, radiologist, or interventional radiologist).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided